CLINICAL TRIAL: NCT00491400
Title: Effect of a Fibrate (Fenofibrate) and a Statin (Atorvastatin) and on Endothelial Dysfunction in Diabetes Mellitus and the Metabolic Syndrome
Brief Title: Effect of a Fibrate and a Statin on Endothelial Dysfunction
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient enrollment
Sponsor: Boston University (Other)
Responsible Party: Principal Investigator, Joseph A. Vita, Professor of Medicine, Boston University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: H-23185
Record Dates: First submitted 2007-06-22; First posted 2007-06-26 (Estimated); Results first posted 2012-10-24 (Estimated); Last update posted 2012-10-24 (Estimated); Status verified 2012-09

CONDITIONS: Diabetes Mellitus; Metabolic Syndrome
Keywords: endothelium; obesity; diabetes mellitus; dyslipidemia
MeSH Terms: conditions — Diabetes Mellitus; Metabolic Syndrome; Obesity; Dyslipidemias | interventions — Fenofibrate; Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fenofibrate First (Active Comparator): Fenofibrate 145 mg/day for 8 weeks First and Atorvastatin 20 mg/day for 8 weeks Second
  Interventions: Drug: Fenofibrate; Drug: Atorvastatin
- Atorvastatin First (Active Comparator): Atorvastatin 20 mg/day for 8 weeks First and Fenofibrate 145 mg/day for 8 weeks Second
  Interventions: Drug: Fenofibrate; Drug: Atorvastatin

INTERVENTIONS:
Drug: Fenofibrate — 140 mg/day for 8 weeks
  Other Names: Tricor
Drug: Atorvastatin — 20 mg/day for 8 weeks
  Other Names: Lipitor

SUMMARY:
The study will compare the effect of atorvastatin to the effect of fenofibrate on endothelial function in patients with diabetes mellitus or the metabolic syndrome.

DETAILED DESCRIPTION:
The study will compare the effect of atorvastatin to the effect of fenofibrate on endothelial function in patients with diabetes mellitus or the metabolic syndrome. The study is a double blind, placebo controlled, crossover study with the order of treatment randomized. Patients will receive each treatment for 8 weeks with a 1 week rest period between treatment periods. Endothelial function will be tested using non-invasive techniques before and after each treatments. A total of 40 subjects with diabetes or the metabolic syndrome will be enrolled at Boston Medical Center.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 30 years
* Adult-onset DM (defined as fasting glucose greater than 125 mg/dl or by ongoing treatment with an oral hypoglycemic agent) or metabolic syndrome (defined as at least 3 of the following: 1. HDL less than 40 mg/dl for men or less than 50 mg/dl for women; 2. triglycerides greater than 150 mg/dl; 3. waist circumference greater than 40 inches for men and greater than 35 inches for women; 4. fasting glucose greater than 100 mg/dl).
* LDL cholesterol level less than 140 mg/dl
* Able to provide informed consent and complete study procedures

Exclusion Criteria:

* Change in therapy for glucose control or blood pressure less than 1 month before entry
* Hemoglobin A1C greater than 8.0%.
* Renal insufficiency (serum creatinine greater than 1.6 mg/dl in men or 1.5 mg/dl in women.
* Any investigational drug less than 1 month before entry.
* Pregnancy (excluded by urine pregnancy test at study entry with ongoing use of reliable form of birth control) or lactation
* Liver function tests or serum creatinine kinase (CK) greater than 3 times upper limit of normal.
* Clinically evident major illnesses or other problem that would make participation inappropriate
* Clinical history of symptomatic cholelithiasis
* Patients with coronary artery disease, peripheral arterial disease, or cerebral vascular disease will not be enrolled if they are currently taking lipid-lowering therapy
* Patients taking more than 40 mg/day of atorvastatin will be excluded. There is no "ceiling" level for patients taking fibrates.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2005-09; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph A Vita, MD, Principal Investigator — Boston University
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients meeting the entry criteria were recruited at Boston Medical Center.
Pre-assignment Details: 101 patients were consented and underwent screening. 73 were excluded because testing demonstrated that they were ineligible. 28 Entered the study 9 withdrew from the study
Groups:
- Fenofibrate First: Participants randomized to receive fenofibrate first and atorvastatin second
- Atorvastatin First: Participants randomized to receive atorvastatin first and fenofibrate second
Period: Overall Study
Arm/Group | Fenofibrate First | Atorvastatin First
Started | 15 | 13
Started First Treatment | 14 (1 withdrew prior to starting fenofibrate) | 13 (None withdrew prior to starting atorvastatin)
Completed First Treatment | 14 (None withdrew during fenofibrate treatment (first treatment)) | 9 (4 withdrew during atorvastatin treatment (first treatment))
Started Second Treatment | 12 (2 withdrew during washout period) | 9 (None withdrew during the washout period)
Finished Second Treatment | 10 (2 withdrew during atorvastatin treatment (second treatment)) | 9 (None withdrew during fenofibrate treatment (second treatment))
Completed | 10 | 9
Not Completed | 5 | 4
Not completed — Withdrawal by Subject | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Fenofibrate First: Fenofibrate First and Atorvastatin Second
- Atorvastatin First: Atorvastatin First and Fenofibrate Second
- Total: Total of all reporting groups
Arm/Group | Fenofibrate First | Atorvastatin First | Total
Number analyzed (Participants) | 15 | 13 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 13 | 28
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 19
  Male | 5 | 4 | 9
Region of Enrollment [Number; unit: participants]
  United States | 15 | 13 | 28

OUTCOME MEASURES:

1. Primary Outcome: Brachial Artery Flow-mediated Dilation
Description: Endothelial function was assessed as brachial artery flow-mediated dilation (FMD) using ultrasound. FMD is calculated as the difference in brachial diameter during hyperemic flow and brachial diameter at baseline divided by brachial diameter at baseline and expressed as percent dilation.
Time Frame: 8 weeks
Population: The number of participants is too few for meaningful analysis.
Groups:
- Fenofibrate Treatment: Effect of fenofibrate on brachial artery FMD
- Atorvastatin Treatment: Effect of atorvastatin on brachial artery FMD
Arm/Group | Fenofibrate Treatment | Atorvastatin Treatment
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Serum Lipids
Description: Effect of the intervention on total cholesterol, HDL, and triglycerides
Time Frame: 8 weeks
Population: Enrollment was insufficient and there are too few subjects for meaningful analysis
Groups:
- Fenofibrate: Effect of fenofibrate treatment on lipid profile
- Atorvastatin: Effect of atorvastatin treatment on lipid profile
Arm/Group | Fenofibrate | Atorvastatin
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Fenofibrate First | Atorvastatin First
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/13
Other Adverse Events (participants affected / at risk) | 0/15 | 0/13

LIMITATIONS AND CAVEATS:
Early termination due to inadequate enrollment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No